CLINICAL TRIAL: NCT02894476
Title: Satisfaction With Care and Quality of Life in Subjects With Substance Dependence
Brief Title: Substance Dependence Satisfaction With Care and Quality Of Life
Acronym: SUBUSQOL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Hospital of Jury-les-Metz, France (Unknown); Healthcare Center of Accompaniment and Prevention in Addictology, Saint-Flour, France (Unknown)
Responsible Party: Sponsor
Other Study IDs: SUBUSQOL
Record Dates: First submitted 2016-08-26; First posted 2016-09-09 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Opiate Dependence; Alcoholism; Early Satisfaction With Substance Dependence Care
Keywords: satisfaction with care; outpatient care; self-reported health status; alcohol dependence; opioid dependence
MeSH Terms: conditions — Opioid-Related Disorders; Alcoholism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The SUBUSQOL cohort aimed to improve knowledge of the quality of ambulatory care, in particular the prognostic role of the early satisfaction with care on the change from baseline quality of self-reported health status in outpatients with alcohol or opioid dependence. It is a multicenter prospective cohort. Satisfaction was assessed using a multidimensional self-administered and validated questionnaire during the early care process. In addition to measuring satisfaction and obtaining sociodemographic and clinical data, this study collected data on the self-reported health status at inclusion and 3, 6 and 12 months after inclusion.

DETAILED DESCRIPTION:
Early satisfaction with care was measured using the quality of care satisfaction questionnaire in outpatient consultation (EQS-C). Data collected during the study included patient sociodemographic, clinical and health status characteristics, as well as physician characteristics. Self-perceived quality of life was assessed using the generic SF-12 and a specific questionnaire in illness disease, the Quality of Life Enjoyment and Satisfaction Questionnaire-Short Form (Q-LES-Q-SF).

ELIGIBILITY:
Inclusion Criteria:

* Outpatients who met the Diagnostic and Statistical Manual, fourth edition (DSM-IV) criteria for alcohol dependence, opioid dependence, or both.
* Patients recruited from the French specialized addiction treatment centers where they began care.
* Patient agreement obtained

Exclusion Criteria:

* Age lower than 18 years
* Inability to complete self-questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients with substance dependence
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2014-04; Primary Completion 2017-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Quality of life score | Change from inclusion at 12 months
  Self-perceived quality of life score using the Short-Form 12 questionnaire (SF-12)
Quality of life score | Change from inclusion at 12 months
  Self-perceived quality of life score using the Quality of life enjoyment and satisfaction questionnaire short form (Q-LES-Q-SF)

SECONDARY OUTCOMES:
Care satisfaction | 15 and 45 days after inclusion
  Outpatient satisfaction score using the quality of care satisfaction questionnaire in outpatient consultation (EQS-C)

CONTACTS AND LOCATIONS:
Overall Officials: Cédric Baumann, PhD, Principal Investigator — CHRU Nancy, PARC
Locations (3):
- France (3):
  - CHS (Hospital of Jury-les-Metz), Jury-les-Metz
  - CSAPA (Healthcare Center of Accompaniment and Prevention in Addictology), University Hospital of Nancy, Nancy
  - ANPAA 15- CSAPA (Healthcare Center of Accompaniment and Prevention in Addictology), Saint-Flour

IPD SHARING:
Plan to Share IPD: No